CLINICAL TRIAL: NCT02485782
Title: Changes in Volumetric Hemodynamic Parameters Induced by Fluid Removal on Hemodialysis
Acronym: CI/HD
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Czyżewski, Łukasz Czyżewski, Medical University of Warsaw
Other Study IDs: C.I/HD/2015/06
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: End Stage Renal Failure on Dialysis; Body Fluid Retention; Impedance; Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hemodialysis patients: * midweek dialysis session
  * patients on maintenance hemodialysis at least 3 months
  * stable dry weight
  * single-pool Kt/V >1.4
  * no clinical cardiovascular disease during the 6 months preceding entry
  Interventions: Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis; Device: BCM- Body Composition Monitor, Fresenius Medical Care; Device: SCHILLER, BR-102 plus, Ambulatory Blood Pressure Monitoring System

INTERVENTIONS:
Device: CardioScreen 1000 - Haemodynamic Measurement System, Medis — Impedance cardiography (ICG)
Device: BCM- Body Composition Monitor, Fresenius Medical Care — Information about the individual fluid status and the nutritional status.
Device: SCHILLER, BR-102 plus, Ambulatory Blood Pressure Monitoring System — Blood pressure monitoring every 15 min during hemodialysis

SUMMARY:
Changes in volumetric hemodynamic parameters and fluid overload (Cardiac Index,Stroke Volume, Thoracic Fluid Content, Systemic Vascular Resistance) were measured using a impedance cardiography (ICG) (CardioScreen 1000 - Haemodynamic Measurement System, Medis. GmbH Ilmenau) beginning 15 min prior to midweek dialysis session and continuous measurement thereafter, with a 15-min period after the termination of hemodialysis. Fluid overload were measured by BCM Monitor Fresenius before hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* patients on maintenance hemodialysis at least 3 months
* stable dry weight
* single-pool Kt/V >1.4
* no clinical cardiovascular disease during the 6 months preceding entry

Exclusion Criteria:

* not meet the above criteria
* episode of illness (for example: infection)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 80 consecutive patients on maintenance hemodialysis were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in volumetric hemodynamic parameter- cardiac index [l/min/m2]) induced by fluid removal on hemodialysis. | 1 day

SECONDARY OUTCOMES:
Changes in volumetric hemodynamic parameter- stroke volume [ml] induced by fluid removal on hemodialysis. | 1 day
Changes in volumetric hemodynamic parameter- systemic vascular resistance [dyn·s·cm-5] induced by fluid removal on hemodialysis. | 1 day
Changes in fluid removal parameter- thoracic fluid content [1/kOhm] during hemodialysis. | 1 day
Changes in blood pressure values [mmHg] induced by fluid removal on hemodialysis. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Wyzgał, Professor, Study Chair — Medical University of Warsaw, Department of Nephrologic Nursing
Locations (1):
- Medical University of Warsaw, Warsaw, Mazovian, Poland

REFERENCES:
- [Background] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Comparative analysis of hypertension and its causes among renal replacement therapy patients. Ann Transplant. 2014 Nov 3;19:556-68. doi: 10.12659/AOT.891248. PMID 25365639
- [Background] Czyzewski L, Wyzgal J, Kolek A. Evaluation of selected risk factors of cardiovascular diseases among patients after kidney transplantation, with particular focus on the role of 24-hour automatic blood pressure measurement in the diagnosis of hypertension: an introductory report. Ann Transplant. 2014 Apr 28;19:188-98. doi: 10.12659/AOT.890189. PMID 24770703
- [Background] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Assessment of health-related quality of life of patients after kidney transplantation in comparison with hemodialysis and peritoneal dialysis. Ann Transplant. 2014 Nov 9;19:576-85. doi: 10.12659/AOT.891265. PMID 25382249